CLINICAL TRIAL: NCT06711276
Title: A Prospective Evaluation of the New Injury Severity Score's Accuracy in Blunt Trauma Patients
Brief Title: Accuracy of the New Injury Severity Score in Evaluating Patients With Blunt Trauma
Acronym: NISS/ER
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241123B
Record Dates: First submitted 2024-11-23; First posted 2024-12-02 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Trauma
Keywords: NISS; Trauma; ER; Death
MeSH Terms: conditions — Wounds and Injuries; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective observational study is to evaluate the predictive utility of the New Injury Severity Score (NISS) in determining mortality outcomes among blunt trauma patients admitted to the Emergency Department of Kadhimiya Educational Hospital, Iraq.

The main questions it aims to answer are:

How accurately does NISS predict mortality in blunt trauma patients? What is the performance of NISS in predicting secondary outcomes, such as the need for intensive care and length of hospital stay?

Participants will:

Be assessed using the NISS score upon their admission to the emergency department.

Have their clinical outcomes, including mortality, need for intensive care, and hospital stay, monitored throughout their hospitalization.

DETAILED DESCRIPTION:
Trauma is the leading cause of death among individuals under 45 years of age, who represent the most productive population of society. According to the World Health Organization, trauma will remain a major driver of years of productive life lost by the end of this decade. Blunt trauma, a common form of injury, typically results in solid organ damage rather than hollow organ injuries.

Trauma management protocols play a vital role in reducing mortality. For example, standardized resuscitation protocols have been shown to decrease mortality by 15% in severely injured patients. The Airway, Breathing, Circulation, Disability, Exposure (ABCDE) approach is a clinically proven framework for managing trauma patients, improving patient outcomes, optimizing team performance, and saving time during life-threatening emergencies. In addition to standardized protocols, scoring systems play a critical role in evaluating the severity of trauma and predicting patient outcomes.

The Injury Severity Score (ISS), introduced in 1974, is one of the most widely used anatomical scoring systems. It evaluates the severity of injuries by dividing the body into six regions: head and neck, face, thorax, abdomen, extremities (including pelvis), and external. Each injury is assigned a score using the Abbreviated Injury Scale (AIS), but only the highest AIS score from each region is used. The ISS is then calculated as the sum of the squares of the top three AIS scores, with a maximum value of 75. Patients with an AIS score of 6 in any region are automatically assigned the maximum ISS score.

However, ISS has limitations. By considering only the most severe injury per body region, which may underestimate the severity of trauma in patients with multiple injuries in the same region. To address this, Osler et al. developed the New Injury Severity Score (NISS) in 1997. Unlike ISS, NISS accounts for the total of squares of the three most severe injuries, regardless of their location in the body, providing a more comprehensive assessment of trauma severity. Studies have shown that NISS often results in higher scores compared to ISS, offering better predictions of patient outcomes in multiple trauma cases.

In addition to anatomical scoring systems like ISS and NISS, physiological scoring systems have been developed to predict outcomes in trauma patients. The Revised Trauma Score (RTS) evaluates physiological parameters, incorporating the Glasgow Coma Scale, systolic blood pressure, and respiratory rate to assess trauma severity and predict mortality.

Research Gap and Study Rationale Although the benefits of NISS over ISS are well-documented globally, there is a lack of localized research evaluating its utility in predicting clinical outcomes in blunt trauma patients in Iraq. Existing studies primarily focus on high-income countries with established healthcare infrastructure, leaving a gap in understanding how such scoring systems perform in resource-limited and post-conflict settings like Iraq.

This study seeks to address this gap by evaluating the predictive accuracy of NISS for blunt trauma patients within Iraq. By assessing the sensitivity, specificity, and overall utility of NISS in the Iraqi healthcare context, this research aims to provide evidence-based recommendations to improve trauma care protocols and patient outcomes. The findings could inform policy development and foster the adoption of standardized trauma assessment tools, thereby strengthening Iraq's healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients admitted to the emergency department, presenting with blunt trauma, such as from motor vehicle accidents, falls, or assaults.
* Patients with adequate documentation of anatomical injuries and physiological parameters required for NISS calculation.
* Injury assessment and NISS calculation completed within the first 6 hours of arrival to ensure accuracy and consistency in trauma evaluation.

Exclusion Criteria:

* Patients under 18 years, pregnant women, or those with pre-existing medical conditions that may alter trauma scoring accuracy or management outcomes.
* Patients presenting with medical emergencies, terminal illnesses, or conditions unrelated to blunt trauma to ensure focus on trauma-specific evaluations.
* Patients declared dead on arrival or who do not receive active treatment in the emergency department.
* Patients or their families refusing participation or withdrawing consent at any stage of the study.
* Patients transferred from or to another facility or those previously treated elsewhere, as this may affect data collection and scoring reliability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of trauma patients presenting to the Emergency Department of Al-Kadhmia Teaching Hospital during the study period. These patients will represent a diverse demographic and clinical profile, including individuals with different injury mechanisms such as motor vehicle accidents, falls, assaults, and sports-related injuries, as well as varying injury severities and outcomes.
  The study will specifically focus on patients for whom the New Injury Severity Score (NISS) can be reliably applied. This includes patients with blunt trauma, where injury severity can be accurately assessed using clinical and radiological data.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 6 days through discharge); Post-Discharge Follow-Up: Day 7, Day 30
  Mortality (death) during hospitalization.
Accuracy Assessment of the New Injury Severity Score (NISS) | the first 6 hours after ER admission
  Range:0 to 75, with higher scores indicating worse outcomes and greater injury severity.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 6 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
Number of Participants Requiring ICU Admission | Up to discharge, an average of 6 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.
The Number of Participants Who Require Surgical Intervention | Up to discharge, an average of 6 days
  need for surgical intervention during a trauma patient's hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Rawa'a A. Sattar A. Wahhab, MBBCH FICS CABMS FACS, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker SP, O'Neill B, Haddon W Jr, Long WB. The injury severity score: a method for describing patients with multiple injuries and evaluating emergency care. J Trauma. 1974 Mar;14(3):187-96. No abstract available. PMID 4814394
- [Background] Thim T, Krarup NH, Grove EL, Rohde CV, Lofgren B. Initial assessment and treatment with the Airway, Breathing, Circulation, Disability, Exposure (ABCDE) approach. Int J Gen Med. 2012;5:117-21. doi: 10.2147/IJGM.S28478. Epub 2012 Jan 31. PMID 22319249
- [Background] van Olden GD, Meeuwis JD, Bolhuis HW, Boxma H, Goris RJ. Advanced trauma life support study: quality of diagnostic and therapeutic procedures. J Trauma. 2004 Aug;57(2):381-4. doi: 10.1097/01.ta.0000096645.13484.e6. PMID 15345989
- [Result] Javali RH, Krishnamoorthy, Patil A, Srinivasarangan M, Suraj, Sriharsha. Comparison of Injury Severity Score, New Injury Severity Score, Revised Trauma Score and Trauma and Injury Severity Score for Mortality Prediction in Elderly Trauma Patients. Indian J Crit Care Med. 2019 Feb;23(2):73-77. doi: 10.5005/jp-journals-10071-23120. PMID 31086450
- [Result] Rapsang AG, Shyam DC. Scoring systems of severity in patients with multiple trauma. Cir Esp. 2015 Apr;93(4):213-21. doi: 10.1016/j.ciresp.2013.12.021. Epub 2014 Jul 8. English, Spanish. PMID 25015031
- [Result] Osler T, Baker SP, Long W. A modification of the injury severity score that both improves accuracy and simplifies scoring. J Trauma. 1997 Dec;43(6):922-5; discussion 925-6. doi: 10.1097/00005373-199712000-00009. PMID 9420106
- [Result] Kuo SCH, Kuo PJ, Chen YC, Chien PC, Hsieh HY, Hsieh CH. Comparison of the new Exponential Injury Severity Score with the Injury Severity Score and the New Injury Severity Score in trauma patients: A cross-sectional study. PLoS One. 2017 Nov 9;12(11):e0187871. doi: 10.1371/journal.pone.0187871. eCollection 2017. PMID 29121653
- [Result] Eid HO, Abu-Zidan FM. New Injury Severity Score is a better predictor of mortality for blunt trauma patients than the Injury Severity Score. World J Surg. 2015 Jan;39(1):165-71. doi: 10.1007/s00268-014-2745-2. PMID 25189444
- [Result] Celso B, Tepas J, Langland-Orban B, Pracht E, Papa L, Lottenberg L, Flint L. A systematic review and meta-analysis comparing outcome of severely injured patients treated in trauma centers following the establishment of trauma systems. J Trauma. 2006 Feb;60(2):371-8; discussion 378. doi: 10.1097/01.ta.0000197916.99629.eb. PMID 16508498
- [Result] Mehta N, Babu S, Venugopal K. An experience with blunt abdominal trauma: evaluation, management and outcome. Clin Pract. 2014 Jun 18;4(2):599. doi: 10.4081/cp.2014.599. eCollection 2014 Jun 18. PMID 25332759
- [Result] van der Vlies CH, Olthof DC, Gaakeer M, Ponsen KJ, van Delden OM, Goslings JC. Changing patterns in diagnostic strategies and the treatment of blunt injury to solid abdominal organs. Int J Emerg Med. 2011 Jul 27;4:47. doi: 10.1186/1865-1380-4-47. PMID 21794108
- See also: Lefering, R. Trauma Score Systems for Quality Assessment. Eur J Trauma 28, 52-63 (2002). — https://doi.org/10.1007/s00068-002-0170-y